CLINICAL TRIAL: NCT03001882
Title: An Exploratory Study of the Biologic Effects and Biomarkers of Nivolumab in Combination With Ipilimumab in Subjects With Treatment-Naive Stage IV or Recurrent Non-Small Cell Lung Cancer (NSCLC)
Brief Title: An Exploratory Study of the Effects of Nivolumab Combined With Ipilimumab in Patients With Treatment-Naive Stage IV or Recurrent Non-Small Cell Lung Cancer (NSCLC)
Acronym: CheckMate 592
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA209-592; 2018-000462-11 (EudraCT Number)
Record Dates: First submitted 2016-12-21; First posted 2016-12-23 (Estimated); Results first posted 2023-06-06 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-04

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Combination therapy (Experimental): Nivolumab + Ipilimumab
  Interventions: Biological: Nivolumab; Biological: Ipilimumab

INTERVENTIONS:
Biological: Nivolumab — Specified dose on specified days
  Other Names: Opdivo; BMS-936558
Biological: Ipilimumab — Specified dose on specified days
  Other Names: Yervoy; BMS-734016

SUMMARY:
The purpose of this study is to explore the possible links between participant characteristics and their cancer, with how effective the combination of nivolumab with ipilimumab is, in participants with Stage IV or recurrent Non-Small Cell Lung Cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, stage IV or recurrent non-small cell lung cancer with no prior systemic anticancer therapy given as primary therapy for advanced or metastatic disease
* Measurable disease by CT or MRI
* Must have full activity or, if limited, must be able to walk and carry out light activities such as light house work or office work

Exclusion Criteria:

* Participants with untreated central nervous system metastases
* Participants with active, known or suspected autoimmune disease
* Prior treatment with any drug that targets T cell co-stimulations pathways (such as checkpoint inhibitors)

Other protocol defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2023-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (35):
- United States (10):
  - Local Institution - 0006, Springdale, Arkansas
  - Local Institution - 0001, New Haven, Connecticut
  - Local Institution - 0005, Jacksonville, Florida
  - Local Institution - 0009, Atlanta, Georgia
  - Local Institution - 0003, St Louis, Missouri
  - Local Institution - 0038, The Bronx, New York
  - Local Institution - 0002, Cleveland, Ohio
  - Local Institution - 0008, Cleveland, Ohio
  - Local Institution - 0007, Greenville, South Carolina
  - Local Institution - 0004, Nashville, Tennessee
- Belgium (5):
  - Local Institution - 0017, La Louvière, Hainaut
  - Local Institution - 0018, Ghent
  - Local Institution - 0028, Ghent
  - Local Institution - 0027, Liège
  - Local Institution - 0016, Sint-Niklaas
- France (4):
  - Local Institution - 0036, Paris
  - Local Institution - 0033, Pierre-Bénite
  - Local Institution - 0034, Strasbourg
  - Local Institution - 0039, Toulon
- Germany (4):
  - Local Institution - 0015, Essen
  - Local Institution - 0014, Immenstadt im Allgäu
  - Local Institution - 0013, Löwenstein
  - Local Institution - 0012, Stuttgart
- Italy (4):
  - Local Institution - 0023, Bergamo
  - Local Institution - 0025, Catania
  - Local Institution - 0026, Parma
  - Local Institution - 0024, Perugia
- Netherlands (2):
  - Local Institution - 0021, Amsterdam
  - Local Institution - 0022, Nijmegen
- Romania (2):
  - Local Institution - 0011, Cluj-Napoca, Cluj
  - Local Institution - 0010, Craiova
- Spain (4):
  - Local Institution - 0031, Barcelona
  - Local Institution - 0029, Madrid
  - Local Institution - 0030, Madrid
  - Local Institution - 0032, Seville

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSStudyConnect.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In Part 1, upon determination of PD-L1 status (cut-off of 1%), 2 cohorts were defined: PD-L1 positive and negative.
  In Part 2, a separate group of participants were treated regardless of their PD-L1 status.
Groups:
- PART 1: PD-L1+ Status; PART 1: PD-L1- Status; PART 1: Not Evaluable/Indeterminate PD-L1 Status; PART 2: PD-L1 Status Independent: Nivolumab + ipilimumab at a flat dose of nivolumab 240 mg as a 30-minute intravenous (IV) infusion every two weeks + ipilimumab 1 mg/kg as a 30-minute IV infusion every 6 weeks. Treatment would continue until disease progression, unacceptable toxicity, withdrawal of consent, the study ending, or a maximum treatment duration of 2 years, whichever occurred first.
Period: Overall Study
Arm/Group | PART 1: PD-L1+ Status | PART 1: PD-L1- Status | PART 1: Not Evaluable/Indeterminate PD-L1 Status | PART 2: PD-L1 Status Independent
Started | 31 | 28 | 1 | 170
Completed (Continuing in treatment period) | 0 | 0 | 0 | 0
Not Completed | 31 | 28 | 1 | 170
Not completed — Death | 1 | 0 | 0 | 3
Not completed — Participant withdrew consent | 0 | 1 | 0 | 5
Not completed — Other reasons | 1 | 2 | 0 | 5
Not completed — Administrative reason by sponsor | 0 | 0 | 0 | 1
Not completed — Participant requested to discontinue study treatment | 0 | 0 | 0 | 2
Not completed — Not reported | 0 | 0 | 0 | 6
Not completed — Maximum clinical benefit | 2 | 3 | 0 | 10
Not completed — AE unrelated to study drug | 3 | 3 | 0 | 11
Not completed — Study Drug Toxicity | 8 | 5 | 0 | 37
Not completed — Disease progression | 16 | 14 | 1 | 90

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PART 1: PD-L1+ Status | PART 1: PD-L1- Status | PART 1: Not Evaluable/Indeterminate PD-L1 Status | PART 2: PD-L1 Status Independent | Total
Number analyzed (Participants) | 31 | 28 | 1 | 170 | 230
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 15 | 0 | 76 | 101
  >=65 years | 21 | 13 | 1 | 94 | 129
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 11 | 0 | 54 | 80
  Male | 16 | 17 | 1 | 116 | 150
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 4 | 6
  Not Hispanic or Latino | 24 | 25 | 1 | 98 | 148
  Unknown or Not Reported | 6 | 2 | 0 | 68 | 76
Race/Ethnicity, Customized [Number; unit: Participants] — Race
  Participants
    White | 27 | 25 | 1 | 164 | 217
    Black or African American | 3 | 3 | 0 | 5 | 11
    Other | 1 | 0 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Per Investigator by Blood TMB (bTMB) Within PD-L1 Subgroup (TMB Cut-point = 16 Mutations/MB)
Description: Objective response rate (ORR) is defined as the percent of treated participants with a best overall response of a complete response (CR) or partial response (PR) assessed by investigator per Response Evaluation Criteria In Solid Tumors (RECIST 1.1).
  PR is at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. CR is disappearance of all target lesions and a reduction in pathological lymph node (whether target or non-target) short axis to <10 mm.
  Blood tumor mutational burden (bTMB) is the total number of nonsynonymous somatic mutations produced by a tumor that are detected in serum.
  CR+PR, confidence interval based on the Clopper and Pearson method.
Time Frame: From first dose up to the date of objectively documented progression, or the date of initiation of palliative local therapy or the date of initiation of subsequent anticancer therapy (up to approximately 58 months)
Population: All treated PD-L1 and bTMB evaluable Part 1 and 2 participants (Blood TMB Cut-point = 16 mutations/MB). Non-evaluable PD-L1 status means that PD-L1 status could not be determined, thus the Arm population did not meet this criteria. Participants in Part 2: PD-L1(+/-) Status groups were stratified from the PART 2: PD-L1 Status Independent Arm. Not all participants were bTMB evaluable. To be analyzed participants had to be both PD-L1 evaluable and bTMB evaluable.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Groups:
- PART 1: PD-L1 + Status; PART 1: PD-L1- Status; PART 1: Not Evaluable/Indeterminate PD-L1 Status; PART 2: PD-L1+ Status; PART 2: PD-L1- Status: Nivolumab + ipilimumab at a flat dose of nivolumab 240 mg as a 30-minute intravenous (IV) infusion every two weeks + ipilimumab 1 mg/kg as a 30-minute IV infusion every 6 weeks. Treatment would continue until disease progression, unacceptable toxicity, withdrawal of consent, the study ending, or a maximum treatment duration of 2 years, whichever occurred first.
Arm/Group | PART 1: PD-L1 + Status | PART 1: PD-L1- Status | PART 1: Not Evaluable/Indeterminate PD-L1 Status | PART 2: PD-L1+ Status | PART 2: PD-L1- Status
Number analyzed (Participants) | 19 | 16 | 0 | 39 | 62
Percent of Participants
  bTMB High (Cut-point = 16-mutations): number analyzed (Participants) | 10 | 10 | 0 | 17 | 33
  bTMB High (Cut-point = 16-mutations) | 30 [6.7 to 65.2] | 50 [18.7 to 81.3] |  | 58.8 [32.9 to 81.6] | 30.3 [15.6 to 48.7]
  bTMB Low (Cut-point = 16-mutations): number analyzed (Participants) | 9 | 6 | 0 | 22 | 29
  bTMB Low (Cut-point = 16-mutations) | 33.3 [7.5 to 70.1] | 33.3 [4.3 to 77.7] |  | 31.8 [13.9 to 54.9] | 24.1 [10.3 to 43.5]

2. Primary Outcome: Objective Response Rate (ORR) Per Investigator by Blood TMB (bTMB) Within PD-L1 Subgroup (Blood TMB Cut-point = 21-mutations/MB)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: All treated PD-L1 and bTMB evaluable Part 1 and Part 2 participants (Blood TMB Cut-point = 21-mutations/MB). Non-evaluable PD-L1 status means that PD-L1 status could not be determined, thus the Arm population did not meet this criteria. Participants in Part 2: PD-L1(+/-) Status groups were stratified from the PART 2: PD-L1 Status Independent Arm. Not all participants were bTMB evaluable. To be analyzed participants had to be both PD-L1 evaluable and bTMB evaluable.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Groups:
- PART 2: PD-L1 + Status; PART 2: PD-L1- Status: Nivolumab + ipilimumab at a flat dose of nivolumab 240 mg as a 30-minute intravenous (IV) infusion every two weeks + ipilimumab 1 mg/kg as a 30-minute IV infusion every 6 weeks. Treatment would continue until disease progression, unacceptable toxicity, withdrawal of consent, the study ending, or a maximum treatment duration of 2 years, whichever occurred first
Arm/Group | PART 1: PD-L1+ Status | PART 1: PD-L1- Status | PART 1: Not Evaluable/Indeterminate PD-L1 Status | PART 2: PD-L1 + Status | PART 2: PD-L1- Status
Number analyzed (Participants) | 19 | 16 | 0 | 39 | 62
Percent of Participants
  bTMB High (Cut-point = 21-mutations): number analyzed (Participants) | 6 | 6 | 0 | 14 | 22
  bTMB High (Cut-point = 21-mutations) | 33.3 [4.3 to 77.7] | 66.7 [22.3 to 95.7] |  | 64.3 [35.1 to 87.2] | 40.9 [20.7 to 63.6]
  bTMB Low (Cut-point = 21-mutations): number analyzed (Participants) | 13 | 10 | 0 | 25 | 40
  bTMB Low (Cut-point = 21-mutations) | 30.8 [9.1 to 61.4] | 30.0 [6.7 to 65.2] |  | 32.0 [14.9 to 53.5] | 20.0 [9.1 to 35.6]

3. Primary Outcome: Objective Response Rate (ORR) Per Investigator by Tissue TMB Within PD-L1 Subgroup (Tissue TMB Cut-point = 10-mutations/MB)
Description: Objective response rate (ORR) is defined as the percent of treated participants with a best overall response of a complete response (CR) or partial response (PR) assessed by investigator per Response Evaluation Criteria In Solid Tumors (RECIST 1.1).
  PR is at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. CR is disappearance of all target lesions and a reduction in pathological lymph node (whether target or non-target) short axis to <10 mm.
  Tissue tumor mutational burden (tTMB) is the total number of nonsynonymous somatic mutations produced by a tumor that are detected in tumor tissue samples.
  CR+PR, confidence interval based on the Clopper and Pearson method.
Time Frame: as for outcome 1
Population: All treated PD-L1 and bTMB evaluable Part 1 and Part 2 participants (Blood TMB Cut-point = 10-mutations/MB). Non-evaluable PD-L1 status means that PD-L1 status could not be determined, thus the Arm population did not meet this criteria. Participants in Part 2: PD-L1(+/-) Status groups were stratified from the PART 2: PD-L1 Status Independent Arm. Not all participants were bTMB evaluable. To be analyzed participants had to be both PD-L1 evaluable and bTMB evaluable.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | PART 1: PD-L1+ Status | PART 1: PD-L1- Status | PART 1: Not Evaluable/Indeterminate PD-L1 Status | PART 2: PD-L1 + Status | PART 2: PD-L1- Status
Number analyzed (Participants) | 19 | 16 | 0 | 31 | 57
Percent of Participants
  tTMB High (Cut-point = 10-mutations): number analyzed (Participants) | 8 | 7 | 0 | 15 | 15
  tTMB High (Cut-point = 10-mutations) | 25.0 [3.2 to 65.1] | 71.4 [29.0 to 96.3] |  | 60.0 [32.3 to 83.7] | 46.7 [21.3 to 73.4]
  tTMB Low (Cut-point = 10-mutations: number analyzed (Participants) | 11 | 9 | 0 | 16 | 42
  tTMB Low (Cut-point = 10-mutations | 27.3 [6.0 to 61.0] | 22.2 [2.8 to 60.0] |  | 25.0 [7.3 to 52.4] | 21.4 [10.3 to 36.8]

4. Secondary Outcome: Objective Response Rate (ORR) for All Treated Participants by Investigator Per RECIST 1.1
Description: Objective response rate (ORR) is defined as the percent of treated participants with a best overall response of a complete response (CR) or partial response (PR) assessed by investigator per Response Evaluation Criteria In Solid Tumors (RECIST 1.1).
  Partial Response (PR) is at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Complete Response (CR) is disappearance of all target lesions and a reduction in pathological lymph node (whether target or non-target) short axis to <10 mm.
  CR+PR, confidence interval based on the Clopper and Pearson method.
Time Frame: From first dose until the date of objectively documented progression, or the date of initiation of palliative local therapy or the date of initiation of subsequent anticancer therapy, whichever occurs first (Up to approximately 67 months)
Population: All treated Part 1 and Part 2 participants
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | PART 1: PD-L1+ Status | PART 1: PD-L1- Status | PART 1: Not Evaluable/Indeterminate PD-L1 Status | PART 2: PD-L1 Status Independent
Number analyzed (Participants) | 31 | 28 | 1 | 170
Percent of Participants | 29.0 [14.2 to 48.0] | 39.3 [21.5 to 59.4] | 0 [0.0 to 97.5] | 29.4 [22.7 to 36.9]

5. Secondary Outcome: Disease Control Rate (DCR) for Part 1
Description: Disease control rate (DCR) is the percent of treated participants with a best overall response of a complete response (CR), partial response (PR), or stable disease (SD), assessed by investigator per Response Evaluation Criteria In Solid Tumors (RECIST 1.1).
  PR is at least a 30% decrease in the sum of diameters of target lesions, using the baseline sum diameters as reference. CR is disappearance of all target lesions and a reduction in short axis to <10 mm of any pathological lymph nodes (target or non-target). SD is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking smallest sum diameters as reference. PD is at least a 20% increase in the sum of diameters of target lesions, taking the smallest sum as reference. The sum must also demonstrate an absolute increase of at least 5 mm. (one or more new lesions is also considered progression). CR+PR, confidence interval based on the Clopper and Pearson method.
Time Frame: as for outcome 4
Population: All treated participants in Part 1. Endpoint pre-specified only for participants treated in Part 1.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | PART 1: PD-L1+ Status | PART 1: PD-L1- Status | PART 1: Not Evaluable/Indeterminate PD-L1 Status
Number analyzed (Participants) | 31 | 28 | 1
Percent of Participants | 58.1 [39.1 to 75.5] | 64.3 [44.1 to 81.4] | 100.0 [2.5 to 100.0]

6. Secondary Outcome: Duration of Response (DOR) for Part 1
Description: DOR is the time between first confirmed response (Complete/Partial Response) and first documented tumor progression (per RECIST 1.1) or death due to any cause. Participants who don't progress or die are censored on the date of their last evaluable tumor assessment. Participants who started subsequent anti-cancer therapy without prior reported progression were censored at the last evaluable tumor assessment prior to or on the date of subsequent anti-cancer therapy.
  PR is at least 30% decrease in the sum of diameters of target lesions, using baseline sum diameters as reference. CR is disappearance of all target lesions and reduction in short axis to <10 mm of any pathological lymph nodes (target or non-target). Progressive Disease (PD) is at least 20% increase in the sum of diameters of target lesions, taking the smallest sum as reference. The sum must also show an overall increase of > 5 mm. (one or more new lesions is also progression). Median computed using Kaplan-Meier method.
Time Frame: From first dose to the date of the first documented tumor progression or death due to any cause (Up to approximately 67 months)
Population: All treated participants in Part 1 who had complete or partial response. Endpoint pre-specified only for participants treated in Part 1.
Measure: Median (Full Range); unit: Months
Arm/Group | PART 1: PD-L1+ Status | PART 1: PD-L1- Status | PART 1: Not Evaluable/Indeterminate PD-L1 Status
Number analyzed (Participants) | 9 | 11 | 0
Months | 24.56 [1.9 to 61.7] | 29.57 [2.8 to 48.9] |

7. Secondary Outcome: Time to Response (TTR) for Part 1
Description: TTR is the time taken from first dosing date to the time the criteria for Complete Response (CR)/Partial Response (PR) are first met.
  Partial Response (PR) is at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Complete Response (CR) is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
Time Frame: From first dose to the time the criteria for Complete Response/Partial Response are first met (Up to approximately 67 months)
Population: as for outcome 6
Measure: Median (Full Range); unit: Months
Arm/Group | PART 1: PD-L1+ Status | PART 1: PD-L1- Status | PART 1: Not Evaluable/Indeterminate PD-L1 Status
Number analyzed (Participants) | 9 | 11 | 0
Months | 1.84 [1.6 to 3.7] | 5.26 [1.7 to 18.5] |

8. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from first dosing date to the date of the first documented tumor progression (per RECIST 1.1) or death due to any cause.
  Participants who neither progress nor die will be censored on the date of their last evaluable tumor assessment. Participants who started any subsequent anti-cancer therapy without a prior reported progression will be censored at the last evaluable tumor assessment prior to or on the date of initiation of subsequent anti-cancer therapy.
  Progressive Disease (PD) is at least a 20% increase in the sum of diameters of target lesions, taking the smallest sum on study as reference. The sum must also show an overall increase of > 5 mm. (one or more new lesions is also progression).
  Median calculated using Kaplan-Meier estimates.
Time Frame: From first dose to the date of the first documented tumor progression or death due to any causes (Assessed up to approximately 67 months)
Population: All treated Part 1 and Part 2 participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | PART 1: PD-L1+ Status | PART 1: PD-L1- Status | PART 1: Not Evaluable/Indeterminate PD-L1 Status | PART 2: PD-L1 Status Independent
Number analyzed (Participants) | 31 | 28 | 1 | 170
Months | 3.71 [1.97 to 8.90] | 4.30 [1.84 to 13.60] | 3.61 [NA to NA] — Insufficient number of participants with events | 6.28 [5.09 to 7.56]

9. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from first dosing date to the date of death. If a participant didn't die, OS will be censored on the last date the participant was known to be alive.
  Median based on Kaplan-Meier estimates.
Time Frame: From first dose to the date of death (Assessed up to approximately 67 months)
Population: All treated Part 1 and Part 2 participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | PART 1: PD-L1+ Status | PART 1: PD-L1- Status | PART 1: Not Evaluable/Indeterminate PD-L1 Status | PART 2: PD-L1 Status Independent
Number analyzed (Participants) | 31 | 28 | 1 | 170
Months | 9.63 [4.47 to 20.57] | 22.29 [11.56 to 25.23] | 9.23 [NA to NA] — Insufficient number of participants with events | 14.78 [11.99 to 20.60]

10. Secondary Outcome: Number of Participants With Adverse Events (AEs) for Study Part 2
Description: An Adverse Event (AE) is any new untoward medical occurrence or worsening preexisting medical condition in a treated participant and that does not necessarily have a causal relationship with treatment.
  An AE can be any unfavorable, unintended sign, symptom, or disease temporally associated with the use of treatment, whether or not related to the treatment.
Time Frame: From first dose to 30 days after last dosing date (assessed up to approximately 27 months)
Population: All treated Part 2 participants. Endpoint pre-specified only for participants treated in Part 2.
Measure: Count of Participants; unit: Participants
Arm/Group | PART 2: PD-L1 Status Independent
Number analyzed (Participants) | 170
Participants | 169

11. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) for Study Part 2
Description: A Serious Adverse Event (SAE) results in death, is life-threatening (defined as an event in which the participant was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe), or requires inpatient hospitalization or causes prolongation of existing hospitalization.
Time Frame: From first dose to 30 days after last dosing date (assessed up to approximately 27 months)
Population: All treated Part 2 participants. Endpoint pre-specified only for participants treated in Part 2.
Measure: Count of Participants; unit: Participants
Arm/Group | PART 2: PD-L1 Status Independent
Number analyzed (Participants) | 170
Participants | 102

12. Secondary Outcome: Number of Participants With Select Adverse Events (AEs) for Study Part 2
Description: as for outcome 10
Time Frame: From first dose to 30 days after last dosing date (up to approximately 27 months)
Population: All treated Part 2 participants. Endpoint pre-specified only for participants treated in Part 2.
Measure: Count of Participants; unit: Participants
Arm/Group | PART 2: PD-L1 Status Independent
Number analyzed (Participants) | 170
Participants
  Gastrointestinal Adverse Events | 68
  Hepatic Adverse Events | 49
  Pulmonary Adverse Events | 17
  Renal Adverse Events | 28
  Skin Adverse Events | 73
  Hypersensitivity/Infusion Reaction | 12

13. Post Hoc Outcome: Extended Collection of Objective Response Rate (ORR) Per Investigator by Blood TMB (bTMB) (TMB Cut-point = 16 Mutations/MB)
Description: as for outcome 1
Time Frame: From first dose up to the date of objectively documented progression, or the date of initiation of palliative local therapy or the date of initiation of subsequent anticancer therapy (up to approximately 67 months)
Population: All treated PD-L1 and bTMB evaluable Part 1 and 2 participants (Blood TMB Cut-point = 16 mutations/MB). Non-evaluable PD-L1 status means that PD-L1 status could not be determined, thus the Arm population did not meet this criteria. Not all participants were bTMB evaluable. To be analyzed participants had to be both PD-L1 evaluable and bTMB evaluable.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Groups:
- PART 1; PART 1: Not Evaluable/Indeterminate PD-L1 Status; PART 2: Nivolumab + ipilimumab at a flat dose of nivolumab 240 mg as a 30-minute intravenous (IV) infusion every two weeks + ipilimumab 1 mg/kg as a 30-minute IV infusion every 6 weeks. Treatment would continue until disease progression, unacceptable toxicity, withdrawal of consent, the study ending, or a maximum treatment duration of 2 years, whichever occurred first.
Arm/Group | PART 1 | PART 1: Not Evaluable/Indeterminate PD-L1 Status | PART 2
Number analyzed (Participants) | 36 | 0 | 131
Percent of Participants
  bTMB High (Cut-point = 16-mutations): number analyzed (Participants) | 20 | 0 | 64
  bTMB High (Cut-point = 16-mutations) | 40.0 [19.1 to 63.9] |  | 34.4 [22.9 to 47.3]
  bTMB Low (Cut-point = 16-mutations): number analyzed (Participants) | 16 | 0 | 67
  bTMB Low (Cut-point = 16-mutations) | 25.0 [7.3 to 52.4] |  | 26.9 [16.8 to 39.1]

14. Post Hoc Outcome: Extended Collection of Objective Response Rate (ORR) Per Investigator by Blood TMB (bTMB) (Blood TMB Cut-point = 21-mutations/MB)
Description: as for outcome 1
Time Frame: as for outcome 13
Population: All treated PD-L1 and bTMB evaluable Part 1 and Part 2 participants (Blood TMB Cut-point = 21-mutations/MB). Non-evaluable PD-L1 status means that PD-L1 status could not be determined, thus the Arm population did not meet this criteria. Not all participants were bTMB evaluable. To be analyzed participants had to be both PD-L1 evaluable and bTMB evaluable.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | PART 1 | PART 1: Not Evaluable/Indeterminate PD-L1 Status | PART 2
Number analyzed (Participants) | 36 | 0 | 131
Percent of Participants
  bTMB High (Cut-point = 21-mutations): number analyzed (Participants) | 12 | 0 | 45
  bTMB High (Cut-point = 21-mutations) | 50.0 [21.1 to 78.9] |  | 44.4 [29.6 to 60.0]
  bTMB Low (Cut-point = 21-mutations): number analyzed (Participants) | 24 | 0 | 86
  bTMB Low (Cut-point = 21-mutations) | 25.0 [9.8 to 46.7] |  | 23.3 [14.8 to 33.6]

15. Post Hoc Outcome: Extended Collection of Objective Response Rate (ORR) Per Investigator by Tissue TMB (Tissue TMB Cut-point = 10-mutations/MB)
Description: as for outcome 3
Time Frame: as for outcome 13
Population: All treated PD-L1 and bTMB evaluable Part 1 and Part 2 participants (Blood TMB Cut-point = 10-mutations/MB). Non-evaluable PD-L1 status means that PD-L1 status could not be determined, thus the Arm population did not meet this criteria. Not all participants were bTMB evaluable. To be analyzed participants had to be both PD-L1 evaluable and bTMB evaluable.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | PART 1 | PART 1: Not Evaluable/Indeterminate PD-L1 Status | PART 2
Number analyzed (Participants) | 35 | 0 | 101
Percent of Participants
  tTMB High (Cut-point = 10-mutations): number analyzed (Participants) | 15 | 0 | 34
  tTMB High (Cut-point = 10-mutations) | 46.7 [21.3 to 73.4] |  | 50.0 [32.4 to 67.6]
  tTMB Low (Cut-point = 10-mutations: number analyzed (Participants) | 20 | 0 | 67
  tTMB Low (Cut-point = 10-mutations | 20.0 [5.7 to 43.7] |  | 19.4 [10.8 to 30.9]

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from their first dose to their study completion (up to approximately 67 months.) SAEs and Other AEs was assessed from first dose to 100 days post the last dose of study therapy (up to approximately an average of 8 months and a maximum of 29 months).
Arm/Group | PART 1: PD-L1+ Status | PART 1: PD-L1- Status | PART 1: Not Evaluable/Indeterminate PD-L1 Status | PART 2: PD-L1 Status Independent
All-Cause Mortality (participants affected / at risk) | 27/31 | 22/28 | 1/1 | 134/170
Serious Adverse Events (participants affected / at risk) | 24/31 | 14/28 | 0/1 | 113/170
Other Adverse Events (participants affected / at risk) | 31/31 | 27/28 | 1/1 | 161/170
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PART 1: PD-L1+ Status (N=31) | PART 1: PD-L1- Status (N=28) | PART 1: Not Evaluable/Indeterminate PD-L1 Status (N=1) | PART 2: PD-L1 Status Independent (N=170)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac tamponade (Cardiac disorders) | 1 | 0 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 1
Nodal rhythm (Cardiac disorders) | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 5
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 3
Hypophysitis (Endocrine disorders) | 0 | 0 | 0 | 4
Thyroiditis (Endocrine disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Autoimmune pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 9
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Adverse drug reaction (General disorders) | 0 | 0 | 0 | 1
Asthenia (General disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 2
Death (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1
General physical health deterioration (General disorders) | 0 | 0 | 0 | 4
Inflammation (General disorders) | 0 | 0 | 0 | 2
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 3
Performance status decreased (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 5
Sudden death (General disorders) | 0 | 0 | 0 | 3
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 0 | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 2
Hepatitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1
Brain abscess (Infections and infestations) | 0 | 0 | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1
Empyema (Infections and infestations) | 0 | 1 | 0 | 0
Encephalitis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1
Klebsiella sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Oral fungal infection (Infections and infestations) | 0 | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 10
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia pneumococcal (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 2
Sepsis (Infections and infestations) | 1 | 0 | 0 | 3
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 2 | 0 | 1
Brachial plexus injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Depressed fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 0 | 0 | 2
Amylase increased (Investigations) | 3 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 2
General physical condition abnormal (Investigations) | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 2 | 0 | 0 | 1
Troponin I increased (Investigations) | 0 | 1 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 5 | 0 | 38
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Phaeochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Encephalitis autoimmune (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0
Metabolic encephalopathy (Nervous system disorders) | 2 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1
Polyneuropathy (Nervous system disorders) | 0 | 0 | 0 | 1
Radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 3
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0
Adnexa uteri mass (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 10
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 6
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0 | 7
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 3
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Embolism (Vascular disorders) | 0 | 1 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PART 1: PD-L1+ Status (N=31) | PART 1: PD-L1- Status (N=28) | PART 1: Not Evaluable/Indeterminate PD-L1 Status (N=1) | PART 2: PD-L1 Status Independent (N=170)
Anaemia (Blood and lymphatic system disorders) | 5 | 6 | 0 | 37
Sinus tachycardia (Cardiac disorders) | 2 | 0 | 0 | 2
Hyperthyroidism (Endocrine disorders) | 1 | 2 | 0 | 16
Hypothyroidism (Endocrine disorders) | 4 | 5 | 0 | 15
Abdominal pain (Gastrointestinal disorders) | 2 | 3 | 0 | 8
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 0 | 7
Colitis (Gastrointestinal disorders) | 0 | 2 | 0 | 4
Constipation (Gastrointestinal disorders) | 6 | 9 | 0 | 25
Diarrhoea (Gastrointestinal disorders) | 7 | 12 | 0 | 65
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 0 | 12
Dyspepsia (Gastrointestinal disorders) | 0 | 4 | 0 | 7
Dysphagia (Gastrointestinal disorders) | 0 | 3 | 0 | 14
Flatulence (Gastrointestinal disorders) | 0 | 2 | 0 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 2 | 0 | 4
Nausea (Gastrointestinal disorders) | 12 | 11 | 0 | 48
Stomatitis (Gastrointestinal disorders) | 1 | 2 | 0 | 8
Vomiting (Gastrointestinal disorders) | 4 | 6 | 0 | 20
Asthenia (General disorders) | 1 | 2 | 0 | 20
Chills (General disorders) | 2 | 2 | 0 | 9
Fatigue (General disorders) | 18 | 16 | 0 | 43
Gait disturbance (General disorders) | 0 | 2 | 0 | 1
Malaise (General disorders) | 2 | 0 | 0 | 4
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 12
Oedema peripheral (General disorders) | 4 | 3 | 0 | 18
Pyrexia (General disorders) | 5 | 5 | 0 | 27
Hypersensitivity (Immune system disorders) | 0 | 2 | 0 | 2
Conjunctivitis (Infections and infestations) | 2 | 0 | 0 | 2
Nasopharyngitis (Infections and infestations) | 2 | 0 | 0 | 9
Sinusitis (Infections and infestations) | 2 | 0 | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 0 | 3 | 0 | 5
Urinary tract infection (Infections and infestations) | 5 | 5 | 0 | 4
Fall (Injury, poisoning and procedural complications) | 2 | 2 | 0 | 5
Alanine aminotransferase increased (Investigations) | 7 | 2 | 0 | 30
Amylase increased (Investigations) | 6 | 5 | 0 | 29
Aspartate aminotransferase increased (Investigations) | 7 | 1 | 0 | 33
Blood alkaline phosphatase increased (Investigations) | 3 | 1 | 0 | 22
Blood bicarbonate decreased (Investigations) | 0 | 2 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 2 | 0 | 1
Blood creatinine increased (Investigations) | 3 | 3 | 0 | 22
International normalised ratio increased (Investigations) | 2 | 0 | 0 | 0
Lipase increased (Investigations) | 6 | 7 | 0 | 28
Platelet count decreased (Investigations) | 2 | 0 | 0 | 4
Weight decreased (Investigations) | 3 | 2 | 0 | 20
White blood cell count decreased (Investigations) | 2 | 0 | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 9 | 9 | 0 | 38
Dehydration (Metabolism and nutrition disorders) | 2 | 3 | 0 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 19
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 5
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 3 | 0 | 12
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 1 | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 4 | 0 | 12
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 3 | 0 | 8
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 4 | 0 | 16
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 3 | 0 | 25
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 2 | 0 | 18
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 7 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 14
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 9
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 0 | 1
Amnesia (Nervous system disorders) | 3 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 5 | 3 | 0 | 12
Dysgeusia (Nervous system disorders) | 0 | 2 | 0 | 8
Headache (Nervous system disorders) | 4 | 5 | 0 | 25
Neuropathy peripheral (Nervous system disorders) | 2 | 1 | 0 | 1
Peroneal nerve palsy (Nervous system disorders) | 0 | 2 | 0 | 0
Anxiety (Psychiatric disorders) | 4 | 0 | 0 | 5
Confusional state (Psychiatric disorders) | 2 | 0 | 0 | 5
Depression (Psychiatric disorders) | 1 | 2 | 0 | 8
Insomnia (Psychiatric disorders) | 2 | 5 | 0 | 12
Acute kidney injury (Renal and urinary disorders) | 1 | 2 | 0 | 3
Haematuria (Renal and urinary disorders) | 0 | 3 | 0 | 3
Pollakiuria (Renal and urinary disorders) | 0 | 4 | 0 | 2
Pelvic pain (Reproductive system and breast disorders) | 2 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 10 | 0 | 45
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 12 | 0 | 45
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 0 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 5
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0 | 8
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 7 | 1 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 0 | 10
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 0 | 17
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 15
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 10 | 1 | 43
Rash (Skin and subcutaneous tissue disorders) | 7 | 8 | 0 | 42
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 6 | 0 | 4
Hot flush (Vascular disorders) | 1 | 2 | 0 | 2
Hypertension (Vascular disorders) | 0 | 5 | 0 | 7
Hypotension (Vascular disorders) | 3 | 4 | 0 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-18): https://cdn.clinicaltrials.gov/large-docs/82/NCT03001882/Prot_SAP_000.pdf